CLINICAL TRIAL: NCT06256822
Title: Effect of Technology-Based Breastfeeding Training After Cesarean on Breastfeeding Success and Self-Efficacy of Mothers
Brief Title: Technology-Based Breastfeeding Training After Cesarean
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Mevlüde Alpaslan Arar, doctor, Ordu University
Other Study IDs: september4
Record Dates: First submitted 2024-01-21; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Cesarean Section; Dehiscence; Breast Feeding; Self Efficacy
Keywords: breastfeeding success; cesarean; education technology; breastfeeding self-efficacy; virtual reality
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim: The aim of this study was to determine the effect of breastfeeding training given with virtual reality (VR) to postpartum primiparous mothers on breastfeeding success and breastfeeding self-efficacy.

Method: The research was designed as a prospective randomized controlled study. In total, 66 women were included in the study, with 31 in the control group and 35 in the intervention group. The intervention group watched a breastfeeding video with VR in the 4th and 24th hours after cesarean. Research data were collected with the sociodemographic information form, LATCH Breastfeeding Charting System and Documentation Tool and the Breastfeeding Self-Efficacy Scale. The study included mothers who gave birth with cesarean section, received breastfeeding counseling during pregnancy, with no vision or hearing disabilities and without any neurological disorder.

ELIGIBILITY:
Inclusion Criteria:

* The study included mothers who gave birth with cesarean section, received breastfeeding counseling during pregnancy, with no vision or hearing disabilities and without any neurological disorder.

Exclusion Criteria:

* Mothers who did not give birth by cesarean section, did not receive breastfeeding counseling during pregnancy, had visual or hearing impairment, or had any neurological disease were not included in the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — breastfeeding mother
Study Population: mothers who gave birth with cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Diagnostic and Assessment Scale | 6 months
  The Latch Breastfeeding Scale was developed by Jensen and Wallace (1993) to objectively diagnose breastfeeding, detect breastfeeding problems, plan breastfeeding education, and create the same language for health professionals. The Cronbach's alpha coefficient of the scale was found to be 0.93. The scale, adapted into Turkish by Yenal and Okumuş (2003), consists of five evaluation steps. LATCH stands for the English expressions of these steps. These evaluation steps are: ''L= Latch on breast'', ''A= Observation of the baby's swallowing movement (Audibleswallowing)'', ''T= Type of nipple'', ''C = The mother's comfort regarding the breast and nipple (Comfort breast/nipple)'', ''H = Holding position of the baby (Hold)''. Items on the scale are scored as 0-1-2. The highest score that can be obtained from the scale is 10 and the lowest score is 0. The Cronbach's alpha coefficient of the scale was found to be 0.95.

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kilic U, Arar M, Oruc MA. The effect of virtual reality on the breastfeeding process: a randomized controlled study. J Perinatol. 2024 Nov;44(11):1611-1616. doi: 10.1038/s41372-024-02077-0. Epub 2024 Jul 31. PMID 39085438